CLINICAL TRIAL: NCT03225092
Title: Efficacy of Platelet-rich Plasma Injections for the Treatment of Persistent Medial Knee Pain After Total Knee Arthroplasty
Brief Title: Platelet-rich Plasma Injections for Persistent Medial Knee Pain After Total Knee Arthroplasty
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit enough study participants
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Baria, Sports Medicine Physician, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0153
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Knee Pain Chronic; Pes Anserinus Bursitis; Status-Post Total Knee Arthroplasty
Keywords: Chronic Knee Pain; Status-Post Total Knee Arthroplasty; Platelet Rich Plasma

STUDY DESIGN:
Intervention Model Description: Observational pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRP Injection (Experimental): Ultrasound-guided platelet rich plasma injection
  Interventions: Biological: Ultrasound-guided platelet rich plasma injection

INTERVENTIONS:
Biological: Ultrasound-guided platelet rich plasma injection — Each participant will receive a single injection into the pes anserine bursa (using the Arthrex Angel system with a setting of 180cc of peripheral blood and 1% hematocrit concentration) under sterile technique

SUMMARY:
This study will investigate the potential effects of platelet rich plasma for the treatment of persistent medial knee pain after total knee arthroplasty. All study participants will receive PRP injections and will be followed up to see if any benefit in regards to pain and/or function is achieved.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of platelet-rich plasma (PRP) injections for the treatment of persistent medial knee pain after total knee arthroplasty (TKA). The investigators hypothesize that PRP injections will provide meaningful pain relief and improved functionality for patients suffering from post-TKA residual pain. The incidence of residual pain after TKA ranges between 10-34%. Many of these patients can be effectively managed by physical therapy, orthotics, and pes anserine bursa corticosteroid injections. However, there remain a number of refractory cases that are frustrating for both the patient and physician. With the advent of interventional pain management, advanced interventions for this clinical problem have focused on selective nerve blocks and ablations targeting the infrapatellar branch of the saphenous nerve. More recently, attention has been paid to the role of patient biology and inflammatory mediators in the development of post-arthroplasty pain (including IL-6 and CRP). If individual patient biology is the foundation of post-TKA pain, then biologic interventions aimed at restoring the balance of these mediators (such as PRP), rather than ablative procedures, seems preferable. Furthermore, while intra-operative PRP has been studied for its effects on wound healing, blood loss, and post-operative pain control, no study has investigated its utility in treating residual medial knee pain after TKA.

All injections will be performed by the same board-certified sports medicine and musculoskeletal ultrasound physician. There will be no activity restrictions following the procedure.

Descriptive statistics will be used to report mean changes in outcome scores. Data will be analyzed with a 2-sample t-test.

ELIGIBILITY:
Inclusion Criteria:

1. Person has had a total knee arthroplasty (total knee replacement)
2. Has experienced persistent medial knee pain beyond six months after surgery
3. Has the presumed diagnosis of pes anserine bursitis
4. No pain relief with conventional treatments such as arch supports (if one is flatfooted), NSAID's, and at least two local steroid injections

Exclusion Criteria:

1. Person has had a prior knee surgical procedure other than the total knee arthroplasty or an arthroscopic debridement procedure
2. Evidence of knee instability, prosthetic loosening, knee infection, radiculopathy, or hip or back pain
3. Personal history of chronic narcotic or recreational drug use, smoking, psychiatric disorders, or a total hip arthroplasty on the same side of the knee arthroplasty
4. Body mass index (BMI) of greater than 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-18 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | Change from baseline to 6 months is primary outcome. Additional outcomes will be collected at 1 and 3 months after procedure.
  Knee Society Scores, a score measurement created by The Knee Society, will be collected as below.

SECONDARY OUTCOMES:
The Hospital for Special Surgery (HSS) Knee Score | Recorded as a baseline and then at 1, 3, and 6 months post intervention
  Knee Scores, a score measurement created by The Hospital for Special Surgery, will be collected as below.
Visual Analog Scale (VAS) for Pain | Recorded as a baseline and then at 1, 3, and 6 months post intervention
  A patient-reported measurement where the subjects will rate their knee pain level by placing a mark along a 100 millimeter line (with each millimeter corresponding to a number, from 0 to 100, 0 meaning no pain at all and 100 meaning the worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baria, MD, MBA, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Shi SM, Meister DW, Graner KC, Ninomiya JT. Selective Denervation for Persistent Knee Pain After Total Knee Arthroplasty: A Report of 50 Cases. J Arthroplasty. 2017 Mar;32(3):968-973. doi: 10.1016/j.arth.2016.09.043. Epub 2016 Oct 8. PMID 27817995
- [Background] Preston S, Petrera M, Kim C, Zywiel MG, Gandhi R. Towards an understanding of the painful total knee: what is the role of patient biology? Curr Rev Musculoskelet Med. 2016 Dec;9(4):388-395. doi: 10.1007/s12178-016-9363-6. PMID 27613710